CLINICAL TRIAL: NCT03286647
Title: Evaluation of Oral Hygiene Self-efficacy in Patients With Grief: a Short-term Randomized Controlled Clinical Trial
Brief Title: Oral Hygiene Self-efficacy in Patients With Grief
Acronym: OHGRIEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Francisco Lotufo Neto, Principal investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 47071315.0.0000.0068
Record Dates: First submitted 2017-08-31; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Grief
Keywords: grief, periodontal disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NORMALGRIEF (Experimental): Oral hygiene instruction
  Interventions: Procedure: Oral hygiene instruction
- COMPLICATEDGRIEF (Experimental): Oral hygiene instruction
  Interventions: Procedure: Oral hygiene instruction
- CONTROLS (Active Comparator): Oral hygiene instruction
  Interventions: Procedure: Oral hygiene instruction

INTERVENTIONS:
Procedure: Oral hygiene instruction — the participants will receive instructions to perform a satisfatory oral hygiene

SUMMARY:
to investigate the effect of oral hygiene self-efficacy in patients with grief (G) and complicated grief (CG)

DETAILED DESCRIPTION:
Aim: to investigate the effect of oral hygiene self-efficacy in patients with grief (G) and complicated grief (CG). Study design: randomized controlled trial. Setting: Institute of Psychiatry-FMUSP (Ipq-FMUSP). Subjects: cases: patients seeking for treatment or under treatment for CG (Group 1), and patients with normal grief (Group 2). Controls: Hospital staff at the HC-FMUSP or volunteers from a list of other studies conducted at the Ipq-FMUSP (Group 3). Method. Psychiatric evaluation: Structured Clinical Interview (SCID), Texas Revised Inventory of Grief (TRIG) and clinical interview. Intervention: instruction of oral hygiene. Dental evaluation: probing depth, clinical attachment level, bleeding on probing, and frequency of plaque at six sites per tooth. Procedures: all participants will complete the psychiatry and dental evaluation at baseline. The bleeding on probing and frequency of plaque will be recorded at baseline, once a week (1 month follow-up) and at 3 months. The probing depth and clinical attachment level will be recorded at baseline and at 3 months. After 3 months, the patients will be referred for dental treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of grief or complicated grief
* Informed consent signature

Exclusion Criteria:

* Patients with severe major depressive disorder at risk for suicide;
* Substance abuse or dependence,
* Psychotic disorders
* Systemic alteration that precludes periodontal clinical examination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-10-05 (Estimated); Primary Completion 2017-10-05 (Estimated); Study Completion 2018-10-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of dental plaque | Change from baseline, 1 and 3 months after oral hygiene instruction
  frequency of dental plaque at 6 sites per tooth

SECONDARY OUTCOMES:
probing depth | Change from baseline and 3 months after oral hygiene instruction
  distance of gingival margin to probe tip
clinical attachment level | Change from baseline and 3 months after oral hygiene instruction
  distance of cemento-enamel junction to probe tip
Bleeding on probing | Change from baseline, 1 and 3 months after oral hygiene instruction
  frequency of bleeding on probing at 6 sites per tooth

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Lotufo-Neto, PhD, Study Chair — Professor; Ana Cristina Solis, PhD, Principal Investigator — Fellowship
Locations (1):
- Department and Institute of Psychiatry - FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No